CLINICAL TRIAL: NCT00304785
Title: Latanoprost Versus Fotil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmaceutical Research Network (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRN 03-026
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2007-10-24 (Estimated); Status verified 2007-10

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

INTERVENTIONS:
Drug: latanoprost 0.005%
Drug: Fotil
Drug: placebo

SUMMARY:
To compare the intraocular pressure effect and safety of latanoprost 0.005% given every evening versus PTFC given twice daily.

ELIGIBILITY:
Inclusion Criteria:

* adults with primary open-angle or pigment dispersion glaucoma, or ocular hypertension
* untreated intraocular pressure should be between 24-36 mm Hg inclusive
* visual acuity should be 5/50 or better in both eyes

Exclusion Criteria:

* presence of exfoliation syndrome or exfoliation glaucoma
* contraindications to study medications
* any anticipated change in systemic hypotensive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-05; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Stewart, MD, Study Director — Pharmaceutical Research Network, LLC; Józef Kałużny, Professor, Principal Investigator — Gabinety Okulistyczne; Krystyna Pecold, Professor, Principal Investigator — Kierownik Kliniki Okulistycznej Akademii Medycznej; Roman Sobecki, Dr. n.med., Principal Investigator — Ordynator Oddziału Okulistycznego Międzyleski Szpital Specjalistyczny; Krystyna Czechowisz-Janicka, Professor, Principal Investigator — Instytut Jaskry; Dariusz Kecik, Professor, Principal Investigator — Katdra Klinika Okulityki Akademii Medycznej w Warszawie
Locations (5):
- Poland (5):
  - Gabinety Okulistyczne, Bydgoszcz
  - Kierownik Kliniki Okulistycznej Akademii Medycznej, Poznan
  - Instytut Jaskry, Warsaw
  - Katdra Klinika Okulityki Akademii Medycznej w Warszawie, Warsaw
  - Ordynator Oddziału Okulistycznego Międzyleski Szpital Specjalistyczny, Warsaw